CLINICAL TRIAL: NCT03416062
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized Trial of the Efficacy and Safety of Remaxol®, a Solution for Infusions Produced by STPF POLYSAN (Russia), in Patients With Malignant Mechanical Jaundice
Brief Title: Remaxol® in Malignant Mechanical Jaundice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REM-CJ-III-16
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Jaundice; Malignant
Keywords: Jaundice, obstructive; Methionine; Succinic acid
MeSH Terms: conditions — Jaundice; Jaundice, Obstructive | interventions — Remaxol; Succinic Acid; Methionine; Inosine; Niacinamide; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remaxol® 400 ml + Placebo 400 ml (Experimental): Treatment with Remaxol® 400 ml IV + Ringer solution 400 ml IV for 10 days. Drug: Remaxol (succinate + methionine + inosine + nicotinamide)
  Interventions: Drug: Remaxol®; Drug: Ringer's Solution
- Remaxol® 800 ml (Experimental): Treatment with Remaxol® 800 ml IV for 10 days. Drug: Remaxol (succinate + methionine + inosine + nicotinamide)
  Interventions: Drug: Remaxol®
- Control (Placebo Comparator): Treatment with Ringer's solution 800 ml IV for 7 days. Drug: Ringer's solution
  Interventions: Drug: Ringer's Solution

INTERVENTIONS:
Drug: Remaxol® — Solution for intravenous infusions, containing succinate, methionine, inosine, and nicotinamide in 400 ml glass bottle
  Other Names: Remaxol (succinate + methionine + inosine + nicotinamide)
  Arms: Remaxol® 400 ml + Placebo 400 ml; Remaxol® 800 ml
Drug: Ringer's Solution — Solution for intravenous infusion, 400 or 800 ml
  Other Names: Placebo
  Arms: Control; Remaxol® 400 ml + Placebo 400 ml

SUMMARY:
The trial intends to study the safety and efficacy of Remaxol® (succinate + methionine + inosine + nicotinamide; POLYSAN Ltd., Russia),solution for infusion for the reduction of hyperbilirubinemia in patients with obstructive jaundice caused by tumor (malignancy).

DETAILED DESCRIPTION:
The study will recruit in-hospital surgical patients with obstructive jaundice caused by malignancies of pancreatic and hepatobiliary zone.

The study consists of the following periods:

* Screening - preliminary examination of patients (duration up to 3 days).
* Period of therapy (including surgery and postoperative period) - treatment with the investigational product Remaxol®, solution for infusions, (NTFF POLYSAN Ltd., Russia) or placebo, as part of standard infusion therapy during the postoperative period of patients with mechanical jaundice of malignant origin (duration 10 days).
* The period of follow-up (duration - 3 weeks after the end of treatment).

After the screening, patients who meet the inclusion criteria and do not have exclusion criteria will be randomly assigned to three groups (1:1:1):

* Group I: treatment with Remaxol® 400 ml IV, and placebo (Ringer solution) 400 ml IV, once a day for 10 days, along with standard infusion therapy.
* Group II: treatment Remaxol® 800 ml IV, once a day for 10 days, along with standard infusion therapy.
* Group III: patients will receive placebo ((Ringer solution) 800 ml IV, once a day for 10 days, along with standard infusion therapy.

Assessment will include physical examination data, vital signs, blood tests (CBC, biochemistry - protein, albumin, AST, ALT, APG, GGTP, LDH, total bilirubin, direct bilirubin, amylase, glucose, electrolytes, creatinine, urea, uric acid, C -reactive protein, lipid profile; coagulogram; urine samples), ECOG assessment, repeated abdominal ultrasound, neurophysiological test for the evaluation of encephalopathy, record of bile volume by drainage (if applicable).

All patients will be followed up for 31 days.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of signed informed consent for participation in the study.
2. Men and women over 18 years of age (incl.).
3. Demonstrated by one or several instrumental methods (ultrasound, cholangiography, CT or MRI) enlargement of intrahepatic bile ducts with visualized obturation of the main bile ducts caused by tumor.
4. Duration of mechanical jaundice less than 30 days, including the first day of the screening period.
5. The status by the classifications Eastern Cooperative Oncology Group (ECOG) scale is 0-2.
6. Life expectancy of more than 3 months.
7. Laboratory data corresponding to the following cutoff limits :

   hemoglobin ≥90 g / l; neutrophils ≥ 1.5x109 / l; Platelets ≥ 75 x 109 / L; AsAT and / or AlAT above 3 х normal but less than 25 х normal Serum creatinine not exceeding 2 × normal, Serum potassium within normal limits
8. Negative urine test for pregnancy in women of reproductive age.
9. For reproductive age: consent to use adequate methods of contraception or for complete abstinence from sexual activity for the period of the study.

Exclusion Criteria:

1. Radical surgery planned within 10 days from the date of randomization.
2. Liver metastases with the biliary block at the level of segmental ducts.
3. Suspicion of metastases in the central nervous system or metastatic arachnoiditis during physical examination; clinically significant ascites.
4. Acute destructive pancreatitis, diffuse peritonitis, ongoing bleeding of any etiology, sepsis (procalcitonin test of 10 ng / ml and above).
5. Liver cirrhosis
6. Presence of clinically significant cardiovascular diseases: chronic cardiac insufficiency III-IV functional class by NYHA, uncontrolled arterial hypertension, acute stroke or acute myocardial infarction in the previous 3 months, unstable angina, uncontrolled arrhythmia and severe heart rhythm disturbances.
7. Pregnancy or lactation.
8. Hypersensitivity to any component of the study drug / placebo and / or intolerance to any component of the study drug / placebo.
9. Regular intake of medications prohibited or not permitted by the study protocol within 4 weeks prior to enrollment or medical indication tio start any medication prohibited or not permitted by the study protocol
10. Concomitant chronic systemic immune or hormonal therapy.
11. Gout.
12. Alcohol and/or drug dependence.
13. Active tuberculosis, HIV infection, syphilis, acute viral hepatitis.
14. Any other conditions / diseases that may interfere with the patient's compliance with the requirements of the Protocol.
15. Mental, physical and other reasons that do not allow the patient to comply with the requirements of the study protocol.
16. Any other significant (by judgement of the investigator) condition that prevents the patient from entering the study.
17. Participation in any clinical trial in the previous 3 months.
18. Staff of the research center and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Time to regression of jaundice | 21 days
  The time (days) from the day of the drainage operation to the reduction of the total bilirubin level down to 90 μmol / l, in experimental (Remaxol®) vs. control (Placebo) groups

SECONDARY OUTCOMES:
Regression of cytolysis (normal alanine aminotransferase and aspartate aminotransferase serum levels) | 11 days
  Proportion of patients in study groups who reached normal serum levels of alanine aminotransferase and aspartate aminotransferase on day 11 from the start of treatment
Regression of cholestasis | 11 days
  Proportion of patients in study groups who reached normal serum levels of alkaline phosphatase, GGTP, total bilirubin, and direct bilirubin on day 11 from the start of treatment
Regression of encephalopathy | 11 days
  Proportion of patients in study groups who had normal brain functioning on day 11, as reflected by the neurophysiological test for the evaluation of the degree of encephalopathy
Serum bilirubin | 21 days
  Dynamics of total and direct bilirubin serum levels against baseline values and between visits in the study groups
Serum alkaline phosphatase | 21 days
  Dynamics of serum alkaline phosphatase level against baseline values and between visits in the study groups
Serum GGTP | 21 days
  Dynamics of serum gamma-glutamyltranspeptidase level against baseline values and between visits in the study groups
Serum alanine aminotransferase | 21 days
  Dynamics of serum alanine aminotransferase level against baseline values and between visits in the study groups
Serum aspartate aminotransferase | 21 days
  Dynamics of serum aspartate aminotransferase level against baseline values and between visits in the study groups
Liver function | 21 days
  State of liver protein synthesis function (as reflected by serum levels of total protein, albumin, INR, PT, PTI, APTT, fibrinogen) against baseline values and/or between visits
Kidney function | 21 days
  State of kidney function (creatinine serum level) against baseline values and/or between visits
Proportion of patients with complications of jaundice | 21 days
  The number of patients in the study groups who developed complications in the postoperative period which were, according to the researcher's assessment, causally related to the obstructive jaundice (for example, purulent cholangitis, sepsis, kidney failure)
Eastern Cooperative Oncology Group (ECOG) Performance Status | 31 days
  Status of patients in the study groups by ECOG (Eastern Cooperative Oncology Group) grades at the end of the study. ECOG Performance Status consists of the following grades:
  0 - fully active, able to carry on all pre-disease performance without restriction;
  1. - restricted but ambulatory and able to carry out work of a light or sedentary nature;
  2. - ambulatory and capable of all selfcare but unable to carry out any work activities;
  3. - capable of only limited selfcare; partially confined to bed or chair;
  4. - completely disabled; cannot carry on any selfcare;
  5. - Dead

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail S. Bogomolov, MD, PhD, Study Director — St. Petersburg State Medical University n.a. I.P.Pavlov
Locations (18):
- Russia (18):
  - GBUZ 'Bryansk City Hospital #1', Bryansk
  - Regional Clinical Hospital of Emergency Care n.a.M.A.Podgorbunsky, Kemerovo
  - KBUZ 'Regional Clinical Hospital', Krasnoyarsk
  - OBUZ 'Kursy Regional Clinical Oncology Dispensary' of Kursky Regional Healthcare Department, Kursk
  - Moscow City Clinical Hospital #1 n.a.N.I.Pirogov, Moscow
  - Moscow City Clinical Hospital #29 n.a.N.A.Bauman, Moscow
  - Omsk Regional Clinical Oncology Center, Omsk
  - GBUZ "Penza Regional Clinical Hospital na N.N.Burdenko", Penza
  - City Clinical Hospital of Emergency Care, Ryazan
  - GBUZ 'Leningrad Regional Oncology Center', Saint Petersburg
  - GBUZ Leningrad Regional Clinical Hospital, Saint Petersburg
  - Hospital for War Veterans, Saint Petersburg
  - North-West State Medical University named after I.I. Mechnikov, Saint Petersburg
  - Saint-Petersburg I.I.Dzanelidze Research Institute of Emergency Medicine, Saint Petersburg
  - SPb GBUZ "City Hospital №26", Saint Petersburg
  - SPb GBUZ 'City Mariinskaya Hospital', Saint Petersburg
  - OGAUZ "Tomsk Regional Clinical Hospital", Tomsk
  - Siberian State Medical University, Tomsk

IPD SHARING:
Plan to Share IPD: No